CLINICAL TRIAL: NCT03013751
Title: A Phase III Extension Study of Udenafil in Adolescents With Single Ventricle Physiology After Fontan Palliation
Brief Title: A Extension Study of Udenafil in Adolescents
Acronym: FUELExten
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mezzion Pharma Co. Ltd (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHN-Udenafil-03; U01HL068270 (NIH)
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Functional Single Ventricle Heart Disease
MeSH Terms: interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug (Experimental): Udenafil administered for 52 weeks
  Interventions: Drug: Udenafil

INTERVENTIONS:
Drug: Udenafil — Active drug

SUMMARY:
This study is a 12-month (52 week) safety extension study to supplement the FUEL Phase III clinical trial to provide safety information regarding the long-term use of udenafil in adolescents with single ventricle congenital heart disease.

DETAILED DESCRIPTION:
This will be an open-label extension study. All enrolled subjects will be provided with udenafil for the duration of the study. Subjects completing the Phase III FUEL study will be eligible for recruitment. Additional subjects will be recruited as needed to ensure a minimum of 300 total subjects enroll. Safety, pharmacodynamic and quality of life data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with Fontan physiology who participated in the FUEL trial or, if they did not participate in FUEL, those who are 12 to less than 19 years of age at enrollment.
2. Participant consent or parental/guardian consent and participant assent.
3. Participant fluent in English, Spanish, or Korean.
4. Current anti-platelet or anticoagulant therapy.

Exclusion Criteria:

1. Height < 132 cm.
2. Weight < 40 kg.
3. Hospitalization for acute decompensated heart failure within the last 12 months.
4. Current intravenous inotropic drugs.
5. Undergoing evaluation for heart transplantation or listed for transplantation.
6. Diagnosis of active protein losing enteropathy or plastic bronchitis within the last three years, or a history of liver cirrhosis.
7. Known Fontan baffle obstruction, branch pulmonary artery stenosis, or pulmonary vein stenosis resulting in a mean gradient of > 4 mm Hg between the regions proximal and distal to the obstruction as measured by either catheterization or echocardiography.
8. Single lung physiology.
9. Maximal VO2 less than 50% of predicted for age and gender at enrollment.
10. Severe ventricular dysfunction assessed qualitatively by clinical echocardiography within six months prior to enrollment.
11. Severe valvar regurgitation, ventricular outflow obstruction, or aortic arch obstruction assessed by clinical echocardiography within six months prior to enrollment.
12. Significant renal, hepatic, gastrointestinal or biliary disorders that could impair absorption, metabolism or excretion of orally administered medications.
13. Inability to complete exercise testing at baseline screening.
14. History of PDE-5 inhibitor use (with the exception of FUEL participation) within 3 months before study onset.
15. Use of any other drug to treat pulmonary hypertension within 3 months before study onset.
16. Known intolerance to oral udenafil.
17. Frequent use of medications or other substances that inhibit or induce CYP3A4.
18. Current use of alpha-blockers or nitrates.
19. Ongoing or planned participation in another research protocol that would either prevent successful completion of planned study testing or invalidate its results.
20. Noncardiac medical, psychiatric, and/or social disorder that would prevent successful completion of planned study testing or would invalidate its results.
21. Cardiac care, ongoing or planned, at a non-study center that would impede study completion.
22. For females: Pregnancy at the time of screening, pregnancy planned before study completion, or refusal to use an acceptable method of contraception for study duration.
23. Unable to abstain or limit intake of grapefruit juice during the duration of the trial.
24. Refusal to provide written informed consent/assent.
25. In the opinion of the primary care physician, the subject is likely to be non-compliant with the study protocol.
26. History of clinically significant thromboembolic event, as adjudicated by study Investigators.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 301 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Paridon, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (24):
- United States (21):
  - Phoenix Children's Hospital/Children's Heart Center at Phoenix Children's Hospital, Phoenix, Arizona
  - Cedars/Sinai Heart Institute, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Cardiac Center/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Heart Institute, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children/Herman B. Wells Center for Pediatric Research, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Congenital Heart Center/C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Mercy Hospital Kansas City, Kansas City, Missouri
  - Washington University St. Louis/St.Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of New York, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Hospital/Dept. of Pediatric Cardiology, Salt Lake City, Utah
  - Seattle Children's Hosptial, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada
- South Korea (2):
  - Sejong General Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Children's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldberg DJ, Zak V, Goldstein BH, McCrindle BW, Menon SC, Schumacher KR, Payne RM, Rhodes J, McHugh KE, Penny DJ, Trachtenberg F, Hamstra MS, Richmond ME, Frommelt PC, Files MD, Yeager JL, Pemberton VL, Stylianou MP, Pearson GD, Paridon SM; Pediatric Heart Network Investigators. Design and rationale of the Fontan Udenafil Exercise Longitudinal (FUEL) trial. Am Heart J. 2018 Jul;201:1-8. doi: 10.1016/j.ahj.2018.03.015. Epub 2018 Apr 3. PMID 29910047

FDAAA 801 VIOLATIONS:
- Issues in Letter Addressed Confirmed — The responsible party has responded, and this matter was resolved administratively. — issued 2026-01-28, released 2025-11-25, posted 2026-02-09
- Violation Identified — Failure to Submit. The entry for this clinical trial was not complete at the time of submission, as required by law. This may or may not have any bearing on the accuracy of the information in the entry. — issued 2025-03-14, released 2020-11-22, posted 2025-04-15

RESULTS

PARTICIPANT FLOW:
Groups:
- In PHN-Udenafil-02 (FUEL) Received Udenafil: Participants in this study arm had received Udenafil in PHN-Udenafil-02 study.
- In PHN-Udenafil-02 (FUEL) Received Placebo: Participants in this study arm had received Placebo in PHN-Udenafil-02 study.
- De novo: Did not participate in PHN-Udenafil-02 study.
Period: Overall Study
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De novo
Started | 128 | 122 | 51
Completed | 128 | 122 | 51
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 128 | 122 | 51 | 301
Age, Customized [Mean (Standard Deviation); unit: Years] — 12 to 18 years old
  Years | 16.1 (2.00) | 16.2 (1.94) | 14.9 (1.89) | 15.9 (2.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 44 | 19 | 118
  Male | 73 | 78 | 32 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 4 | 35
  Not Hispanic or Latino | 110 | 107 | 47 | 264
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 2 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 6 | 14
  White | 119 | 107 | 38 | 264
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 2 | 6 | 2 | 10
Weight [Mean (Standard Deviation); unit: kilogram] | 59.2 (13.62) | 60.7 (13.58) | 57.7 (15.10) | 59.5 (13.86)
Height [Mean (Standard Deviation); unit: centimeter] | 164.2 (10.18) | 166.3 (8.84) | 163.2 (9.08) | 164.9 (9.52)
Maximal VO2 [Mean (Standard Deviation); unit: mL/min] — Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points). VO2 has been presented in mL/min (i.e., not adjusted for body weight).
  mL/min
    number analyzed (Participants) | 90 | 93 | 12 | 195
    (all) | 1607.3 (470.80) | 1637.6 (444.26) | 1421.7 (261.32) | 1610.4 (449.13)
Myocardial Performance Index (MPI) [Mean (Standard Deviation); unit: Ratio] — The MPI is a measure of systolic and diastolic function determined by velocities from blood pool Doppler assessment of the inflow and outflow tract of the dominant ventricle. MPI is calculated by dividing the sum of the isovolumetric contraction and relaxation time by the ejection time at each site measurement. The MPI is used to measure global cardiac dysfunction; decreases in MPI correspond with improved cardiac function and increases in MPI correspond with diminished cardiac function. The mean MPI in healthy people without heart disease is approximately 0.35. Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points).
  Ratio
    number analyzed (Participants) | 59 | 60 | 4 | 123
    (all) | 0.43 (0.118) | 0.46 (0.152) | 0.59 (0.326) | 0.45 (0.146)
Log-transformed Reactive Hyperemia Index (lnRHI) [Mean (Standard Deviation); unit: Natural log-transformed RHI (lnRHI)] — The Reactive Hyperemia Index (RHI) is the ratio of the amount of blood flow after the release of a period of vessel occlusion relative to baseline amount of blood flow. Because the amount of blood does not decrease after release of vessel occlusion, the minimum value for the RHI is 1.0, which would indicate no change in blood flow. There is no upper limit for this ratio, and higher values are generally thought to represent a healthier endothelial response. In this study, as in other studies, we used the natural log of RHI (lnRHI) to normalize the data. Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points).
  Natural log-transformed RHI (lnRHI)
    number analyzed (Participants) | 82 | 83 | 8 | 173
    (all) | 1.748 (0.4940) | 1.757 (0.5403) | 1.585 (0.3987) | 1.745 (0.5117)
Serum BNP [Mean (Standard Deviation); unit: pg/mL] — Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points).
  pg/mL
    number analyzed (Participants) | 48 | 53 | 0 | 101
    (all) | 18.25 (14.796) | 15.58 (18.638) |  | 16.85 (16.891)
Pediatric Quality of Life (PedsQL)-Physical Functioning-Child reported [Mean (Standard Deviation); unit: score on a scale] — The Pediatric Quality of Life Inventory (PedsQL) - Physical Function Scale is calculated from a child's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better reported physical function. Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points).
  score on a scale
    number analyzed (Participants) | 111 | 119 | 37 | 267
    (all) | 73.68 (13.845) | 74.40 (16.142) | 73.99 (13.722) | 74.04 (14.848)
Pediatric Quality of Life (PedsQL)-Physical Functioning-Parent reported [Mean (Standard Deviation); unit: score on a scale] — The Pediatric Quality of Life Inventory (PedsQL) - Physical Function Scale is calculated from parent's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better reported physical function. Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points).
  score on a scale
    number analyzed (Participants) | 106 | 106 | 35 | 247
    (all) | 76.43 (17.064) | 76.90 (14.948) | 73.24 (18.112) | 76.18 (16.324)
Pediatric Quality of Life (PedsQL)-Psychosocial Health Summary Score-Child reported [Mean (Standard Deviation); unit: score on a scale] — The Pediatric Quality of Life Inventory (PedsQL) - Psychosocial Health Summary Scale is calculated from a child's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better reported psychosocial health. Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points).
  score on a scale
    number analyzed (Participants) | 111 | 119 | 37 | 267
    (all) | 73.40 (14.562) | 73.11 (16.306) | 70.23 (14.429) | 72.83 (15.327)
Pediatric Quality of Life (PedsQL)-Psychosocial Health Summary Score-Parent reported [Mean (Standard Deviation); unit: score on a scale] — The Pediatric Quality of Life Inventory (PedsQL) - Psychosocial Health Summary Scale is calculated from parent's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better reported psychosocial health. Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points).
  score on a scale
    number analyzed (Participants) | 106 | 106 | 35 | 247
    (all) | 70.40 (17.258) | 73.64 (16.558) | 65.50 (17.458) | 71.10 (17.139)
Pediatric Quality of Life (PedsQL)-Functional Health Status Score-Child reported [Mean (Standard Deviation); unit: score on a scale] — The Pediatric Quality of Life Inventory (PedsQL) - Functional Health Status Score is calculated from a child's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better functional health status. Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points).
  score on a scale
    number analyzed (Participants) | 111 | 119 | 37 | 267
    (all) | 73.50 (13.108) | 73.56 (14.755) | 71.53 (12.802) | 73.26 (13.795)
Pediatric Quality of Life (PedsQL)-Functional Health Status Score-Parent reported [Mean (Standard Deviation); unit: score on a scale] — The Pediatric Quality of Life Inventory (PedsQL) - Functional Health Status Score is calculated from parent's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better functional health status. Population: Baseline results only presented for subjects who have data at 52 weeks (i.e., paired-data points).
  score on a scale
    number analyzed (Participants) | 106 | 106 | 35 | 247
    (all) | 72.49 (15.621) | 74.75 (14.248) | 68.20 (15.488) | 72.85 (15.122)

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Emergent Adverse Events
Description: Summary of Treatment Emergent Adverse Events
Time Frame: 52 Weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Total: Total number of subjects who participated in FUEL open label extension study.
Arm/Group | Total
Number analyzed (Participants) | 301
Participants
  Subjects with one or more TEAEs adverse event (TEAE) | 257
  Subjects with one or more drug-related TEAEs | 206
  Subjects with one or more TEAEs of Grade >=3 | 31
  Subjects with one or more SAEs | 54
  Subjects with one or more drug-related SAEs | 15
  Subjects who temporarily stopped study drug for one or more TEAEs | 35
  Subjects who permanently discontinued study drug for one or more TEAEs | 21

2. Secondary Outcome: Change in Maximal VO2
Description: Change in Maximal VO2 from baseline to 52 weeks
Time Frame: 52 Weeks
Population: Results presented only for subjects who have data at baseline and 52 weeks (i.e., paired-data points). VO2 has been presented in mL/min (i.e., not adjusted for body weight).
Measure: Mean (Standard Deviation); unit: mL/min
Groups:
- In PHN-Udenafil-02 (FUEL) Received Udenafil: Subjects received 26 weeks of udenafil in the double-blind trial (FUEL) and then received 52 weeks of udenafil in the open-label trial.
- In PHN-Udenafil-02 (FUEL) Received Placebo: Subjects received 26 weeks of placebo in the double-blind trial (FUEL) and then received 52 weeks of udenafil in the open-label trial.
- De Novo: Subjects not in the FUEL trial but joined the open-label trial de novo and received 52 weeks of udenafil.
- Total: Total number of subjects who participated in the open-label extension study
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 90 | 93 | 12 | 195
mL/min
  Baseline | 1607.3 (470.80) | 1637.6 (444.26) | 1421.7 (261.32) | 1610.4 (449.13)
  52 weeks | 1646.1 (433.94) | 1703.0 (434.31) | 1425.0 (269.12) | 1659.6 (429.34)

3. Secondary Outcome: Change in Log-transformed Reactive Hyperemia Index (lnRHI)
Description: Change from baseline to 52 weeks in Log-transformed Reactive Hyperemia Index (lnRHI). The Reactive Hyperemia Index (RHI) is the ratio of the amount of blood flow after the release of a period of vessel occlusion relative to baseline amount of blood flow. Because the amount of blood does not decrease after release of vessel occlusion, the minimum value for the RHI is 1.0, which would indicate no change in blood flow. There is no upper limit for this ratio, and higher values are generally thought to represent a healthier endothelial response. In this study, as in other studies, we used the natural log of RHI (lnRHI) to normalize the data.
Time Frame: 52 Weeks
Population: Results presented only for subjects who have data at baseline and 52 weeks (i.e., paired-data points).
Measure: Mean (Standard Deviation); unit: Natural log-transformed RHI (lnRHI)
Groups:
- De Novo: Subjects who did not participate in the FUEL trial but joined the open-label trial de novo and received 52 weeks of udenafil.
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 82 | 83 | 8 | 173
Natural log-transformed RHI (lnRHI)
  Baseline | 1.748 (0.4940) | 1.757 (0.5403) | 1.585 (0.3987) | 1.745 (0.5117)
  52 weeks | 1.759 (0.5171) | 2.037 (0.6405) | 1.960 (0.5315) | 1.902 (0.5931)

4. Secondary Outcome: Change in Serum BNP
Description: Change in Serum BNP from baseline to 52 weeks
Time Frame: 52 Weeks
Population: Results presented only for subjects who have data at baseline and 52 weeks (i.e., paired-data points). The de novo population did not have any paired-data.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 48 | 53 | 0 | 101
pg/mL
  Baseline | 18.25 (14.796) | 15.58 (18.638) |  | 16.85 (16.891)
  52 weeks | 26.18 (24.241) | 23.13 (24.584) |  | 24.58 (24.347)

5. Secondary Outcome: Change in Myocardial Performance Index (MPI)
Description: Change in Myocardial Performance Index from baseline to 52 weeks
Time Frame: 52 Weeks
Population: Efficacy population
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 59 | 60 | 4 | 123
mL/min
  Baseline | 0.43 (0.118) | 0.46 (0.152) | 0.59 (0.326) | 0.45 (0.146)
  52 weeks | 0.43 (0.140) | 0.41 (0.140) | 0.53 (0.148) | 0.42 (0.141)

6. Secondary Outcome: Change in PedsQL Physical Functioning (Child Reported)
Description: Change in PedsQL Physical Functioning (Child Reported) from baseline to 52 weeks. The Pediatric Quality of Life Inventory (PedsQL) - Physical Function Scale is calculated from a child's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better reported physical function.
Time Frame: 52 Weeks
Population: Results presented only for subjects who have data at baseline and 52 weeks (i.e., paired-data points).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 111 | 119 | 37 | 267
score on a scale
  Baseline | 73.68 (13.845) | 74.40 (16.142) | 73.99 (13.722) | 74.04 (14.848)
  52 weeks | 74.75 (15.823) | 74.10 (17.691) | 73.56 (14.669) | 74.30 (16.482)

7. Secondary Outcome: Change in PedsQL Physical Functioning (Parent Reported)
Description: Change in PedsQL Physical Functioning (Parent Reported) from baseline to 52 weeks. The Pediatric Quality of Life Inventory (PedsQL) - Physical Function Scale is calculated from parent's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better reported physical function.
Time Frame: 52 Weeks
Population: Results presented only for subjects who have data at baseline and 52 weeks (i.e., paired-data points).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 106 | 106 | 35 | 247
score on a scale
  Baseline | 76.43 (17.064) | 76.90 (14.948) | 73.24 (18.112) | 76.18 (16.324)
  52 weeks | 75.99 (18.205) | 76.10 (15.772) | 74.11 (13.946) | 75.77 (16.582)

8. Secondary Outcome: Change in PedsQL Psychosocial Health Summary Score (Child Reported)
Description: Change in PedsQL Psychosocial Health Summary Score (Child reported) from baseline to 52 weeks. The Pediatric Quality of Life Inventory (PedsQL) - Psychosocial Health Summary Scale is calculated from a child's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better reported psychosocial health.
Time Frame: 52 Weeks
Population: Results presented only for subjects who have data at baseline and 52 weeks (i.e., paired-data points).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 111 | 119 | 37 | 267
score on a scale
  Baseline | 73.40 (14.562) | 73.11 (16.306) | 70.23 (14.429) | 72.83 (15.327)
  52 weeks | 73.01 (17.451) | 72.37 (17.174) | 71.31 (17.015) | 72.49 (17.212)

9. Secondary Outcome: Change in PedsQL Psychosocial Health Summary Score (Parent Reported)
Description: Change in PedsQL Psychosocial Health Summary Score (Parent reported) from baseline to 52 weeks. The Pediatric Quality of Life Inventory (PedsQL) - Psychosocial Health Summary Scale is calculated from parent's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better reported psychosocial health.
Time Frame: 52 Weeks
Population: Results presented only for subjects who have data at baseline and 52 weeks (i.e., paired-data points).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 106 | 106 | 35 | 247
score on a scale
  Baseline | 70.40 (17.258) | 73.64 (16.558) | 65.50 (17.458) | 71.10 (17.139)
  52 weeks | 71.18 (18.027) | 72.32 (17.099) | 68.24 (14.730) | 71.25 (17.184)

10. Secondary Outcome: Change in PedsQL Functional Health Status Score (Child Reported)
Description: Change in PedsQL Functional Health Status Score (Child reported) from baseline to 52 weeks. The Pediatric Quality of Life Inventory (PedsQL) - Functional Health Status Score is calculated from a child's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better functional health status.
Time Frame: 52 Weeks
Population: Results presented only for subjects who have data at baseline and 52 weeks (i.e., paired-data points).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 111 | 119 | 37 | 267
score on a scale
  Baseline | 73.50 (13.108) | 73.56 (14.755) | 71.53 (12.802) | 73.26 (13.795)
  52 weeks | 73.64 (15.794) | 72.98 (15.735) | 72.09 (14.762) | 73.13 (15.580)

11. Secondary Outcome: Change in PedsQL Functional Health Status Score (Parent Reported)
Description: Change in PedsQL Functional Health Status Score (Parent reported) from baseline to 52 weeks. The Pediatric Quality of Life Inventory (PedsQL) - Functional Health Status Score is calculated from parent's answers to a short questionnaire. The range of possible scores is 0-100, and higher scores indicate better functional health status.
Time Frame: 52 Weeks
Population: Results presented only for subjects who have data at baseline and 52 weeks (i.e., paired-data points).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In PHN-Udenafil-02 (FUEL) Received Udenafil | In PHN-Udenafil-02 (FUEL) Received Placebo | De Novo | Total
Number analyzed (Participants) | 106 | 106 | 35 | 247
score on a scale
  Baseline | 72.49 (15.621) | 74.75 (14.248) | 68.20 (15.488) | 72.85 (15.122)
  52 weeks | 72.85 (16.638) | 73.63 (15.044) | 70.28 (13.181) | 72.82 (15.491)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Subjects taking the study drug for 52 weeks
Groups:
- Total: Total number of subjects who participated in the open-label extension study (PHN-Udenafil-03)
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 0/301
Serious Adverse Events (participants affected / at risk) | 54/301
Other Adverse Events (participants affected / at risk) | 257/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=301)
Anaemia (Blood and lymphatic system disorders) | 2
Cardiac Failure (Cardiac disorders) | 4
Supraventricular tachycardia (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 2
Atrial flutter (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Blindness transient (Eye disorders) | 1
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Tooth Impacted (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Exercise tolerance decreased (General disorders) | 1
Oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Cardiac cirrhosis (Hepatobiliary disorders) | 1
Congestive hepatopathy (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Coronavirus infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Burkitt's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transient ischaemic attack (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Device malfunction (Product Issues) | 1
Depression (Psychiatric disorders) | 3
Suicide attempt (Psychiatric disorders) | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Intentional self injury (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Angioplasty (Surgical and medical procedures) | 1
Scoliosis surgery (Surgical and medical procedures) | 1
Tympanoplasty (Surgical and medical procedures) | 1
Hyptension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=301)
Headache (Nervous system disorders) | 122
Flushing (Vascular disorders) | 52
Dizziness (Nervous system disorders) | 42
Nasopharyngitis (Infections and infestations) | 41
Chest pain (General disorders) | 35
Fatigue (General disorders) | 31
Nausea (Gastrointestinal disorders) | 31
Upper respiratory tract infection (Infections and infestations) | 31
Migraine (Nervous system disorders) | 25
Influenza (Infections and infestations) | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Pyrexia (General disorders) | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21
Sinusitis (Infections and infestations) | 21
Vomiting (Gastrointestinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20
Abdominal pain upper (Gastrointestinal disorders) | 18
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18
Pharyngitis streptococcal (Infections and infestations) | 17
Ear infection (Infections and infestations) | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16
Palpitations (Cardiac disorders) | 16
Depression (Psychiatric disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT03013751/Prot_SAP_000.pdf